CLINICAL TRIAL: NCT05900856
Title: Effect of Ultrasound Cavitation on Static and Dynamic Balance in Obese Postnatal Women With Diastasis Recti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Maher Ahmed Zahran, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p. t.REC/012/003570
Record Dates: First submitted 2023-05-26; First posted 2023-06-13 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Rectus Diastasis
Keywords: Ultrasound Cavitation, Static Balance, Dynamic Balance

STUDY DESIGN:
Intervention Model Description: ultrasound cavitation and low caloric diet regimen
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low caloric diet regimn (Experimental): patients will follow low caloric diet regimn (1600: 2000 Kcal/ day), lipids approximately (20: 35%) of total caloric intake, protein approximately (10: 35%) of total caloric intake and high complexed carbohydrate intake approximately (45: 65%) of total caloric intake (with increased fiber-rich whole grain breads, cereals, fruits and vegetables), for eight weeks.
  Interventions: Other: low caloric diet regimen
- ultrasound cavitation for 30 minutes, twice per week for eight weeks and low caloric diet regimn (Experimental): ultrasound cavitation, Dae Yang, Mabel 6, frequency (50: 60) Hz, power consumption 150 W, power input AC (100: 230) V, hand probe diameter 8.0 cm, serial number DY73-15037, produced by DAEYANG MEDICAL company, made in Korea. the device will be applied for 30 minutes on the abdominal area, twice per week for eight weeks.
  low caloric diet regimn patients will follow low caloric diet regimn (1600: 2000 Kcal/ day), lipids approximately (20: 35%) of total caloric intake, protein approximately (10: 35%) of total caloric intake and high complexed carbohydrate intake approximately (45: 65%) of total caloric intake (with increased fiber-rich whole grain breads, cereals, fruits and vegetables), for eight weeks.
  Interventions: Other: low caloric diet regimen; Device: ultrasound cavitation

INTERVENTIONS:
Other: low caloric diet regimen — lipids approximately (20: 35%) of total caloric intake, protein approximately (10: 35%) of total caloric intake and high complexed carbohydrate intake approximately (45: 65%) of total caloric intake (with increased fiber-rich whole grain breads, cereals, fruits and vegetables), for eight weeks.
  Other Names: hypocaloric diet (1600: 2000 Kcal/ day)
Device: ultrasound cavitation — patients will assume standing position, the abdominal area will be divided vertically into 2 equal sections, right and left segment, extending bilaterally from the line stretching between the mid axilla above and the iliac crest below, and upward from center of diaphragm to the midpoint extending between two iliac crest below, then from supine lying position the cavitation head will be applied on each abdominal segment for 15 minutes with total treatment time 30 minutes twice per week for eight weeks
  Other Names: Dae Yang, Mabel 6, serial number DY73-15037, produced by DAEYANG MEDICAL company
  Arms: ultrasound cavitation for 30 minutes, twice per week for eight weeks and low caloric diet regimn

SUMMARY:
the aim of this study is to investigate the efficacy of ultrasound cavitation on static and dynamic balance in obese postnatal women with diastasis recti

DETAILED DESCRIPTION:
Rectus diastasis defined as the widening of the linea alba by more than 2 cm at the midline. A great proportion of pregnant women are complaining from rectus diastasis during pregnancy reaching 100% of all women that may continue for years after delivery in 66% of women, and do not return to the first state automatically. This occurs due to a combination of physiologic, hormonal and mechanical factors, leading to reduction of abdominal muscle functional strength, increased low back pain out of increased lumbar hyperlordosis and postural instability, which may seriously disable woman from taking care of her baby, perform her daily activities. Weight gain is one of the predisposing factors that increases the possibility of developing rectus diastasis postpartum. Being obese increases liability to have rectus diastasis as carrying excess abdominal fats puts greater pressure against linea alba and can develop or aggravate symptoms for both men and women. This massively displaces the center of gravity anteriorly, disturbs body balance, increases joint loads and influences negatively pelvis posture leading to increased anterior pelvic tilt with subsequent exaggerated lumbar hyperlordosis. Ultrasound cavitation is the most revolutionary method that destroys excess body fat through creating microbubbles and releasing energy that breaks down fat cells. This trial has two groups: one will be treated by low caloric diet regimen only and the second one will be treated by ultrasound cavitation in addition to low caloric diet regimen for eight weeks

ELIGIBILITY:
Inclusion Criteria:

1. All women had a diastasis recti more than 2.5 cm and less than 4 cm in supra umbilical region.
2. Their ages were ranged from 25: 35 years.
3. Their BMI was more than 30 Kg/ m2.
4. All women were with lumbar hyperlordosis.
5. All women were multipara.
6. Their mode of delivery was normal vaginal delivery.
7. They were selected from 2: 5 months postnatal.

Exclusion Criteria:

1. Previous cesarean section.
2. Previous abdominal and/ or back operation.
3. Spinal disorders.
4. Abdominal skin diseases.
5. Serious diseases such as heart disease, pace maker, uncontrolled diabetes or hypertension, autoimmune disease, malignancy, gastric ulcer, liver or renal failure and any other contraindication for body sculpting-weight loss.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — obese postnatal women with rectus diastasis
Enrollment: 60 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Static postural balance | up to eight weeks
  The Biodex Balance System SD (model: TP-3040-15, DC input: 19V-6.32A, connected to computer software version 4.0.06, 2017, serial number: R712010010, made in Taiwan) will be used to measure overall stability index of static postural balance for all patients
Dynamic postural balance | up to eight weeks
  The Biodex Balance System SD (model: TP-3040-15, DC input: 19V-6.32A, connected to computer software version 4.0.06, 2017, serial number: R712010010, made in Taiwan) will be used to measure overall stability index of dynamic postural balance for all patients

SECONDARY OUTCOMES:
Abdominal subcutaneous fat thickness | up to eight weeks
  Ultrasound imaging unit (Mindary DP10, linear probe, with 10 MHz frequency, serial number: bn- 75013216, made in China) will be used to measure abdominal subcutaneous fat thickness at the umbilical level from supine lying position for all patients
Inter recti distance | up to eight weeks
  Ultrasound imaging unit (Mindary DP10, convex probe, with 5 MHz frequency, serial number: bn- 75013216, made in China) will be used to measure resting inter recti distance 2.5 cm above the upper margin of umbilicus from crock lying position for all patients
Lumbar lordotic angle | up to eight weeks
  Spinal mouse (MEDIMOUSE) IDIAG M360 pro, pc-Software, 7.4.0., serial number: *112D2A24*, made in Switzerland) will be used to measure lumbar lordotic angle from standing position

CONTACTS AND LOCATIONS:
Locations (1):
- Asmaa Maher Ahmed Zahran, Giza, Egypt